CLINICAL TRIAL: NCT04658433
Title: The Effect of Omega -3 Supplements on the Serum Levels of ACE/ACE2 Ratio as a Potential Key in Cardiovascular Disease and COVID-19; A Randomized Clinical Trial in the COVID-19 Uninfected Jordanian People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science Private University (Other)
Responsible Party: Principal Investigator, Mahmoud Suleiman Abu-Samak, Mahmoud S Abu-Samak, PhD Study Principal Investigator Department of Clinical Pharmacy and Therapeutics, Applied Science Private University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-PHA-22
Record Dates: First submitted 2020-12-05; First posted 2020-12-08 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Cardiovascular Risk Factor; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- n-3FA group (Experimental): Dietary Supplement: 1,000 mg of wild salmon and fish oil complex once daily, which contains 300 mg of omega3-FA for 8 weeks.
  Interventions: Dietary Supplement: 300 mg of omega3-FA
- Control group (No Intervention)

INTERVENTIONS:
Dietary Supplement: 300 mg of omega3-FA — The participant will receive 1,000 mg of wild salmon and fish oil complex once daily, which contains 300 mg of omega3-FA.
  Arms: n-3FA group

SUMMARY:
The Renin-Angiotensin-Aldosterone System (RAAS) is involved in blood pressure regulation and electrolyte balance. Angiotensin-converting enzyme (ACE) is a critical regulator of RAAS by cleaving angiotensin (Ang1) to Angiotensin2 (Ang2), which is the most powerful biologically active product of RAAS [1]. In the same context, angiotensin-converting enzyme 2 (ACE2) converts Ang2 to Ang (1-7), which is a vasodilator, antithrombotic, and antihypertrophic peptide [2]. ACE2 which is found in many tissues [3] has opposite effects to ACE on the heart, kidneys, and lungs [4]. Many pathological conditions, in particular cardiovascular disease (CVD), have shown a link between a disturbance in ACE/ACE2 ratio and the downregulation of ACE2 levels [5]. Also, ACE/ACE2 has been reported to be higher in moderate to severe chronic heart failure [6] as well as systolic blood pressure [7]. Recently, an elevated ACE/ACE2 ratio is linked to Coronavirus disease 2019 (COVID-19). SARS-COV2 enters target cells by binding of the spike protein to ACE2 and a specific transmembrane serine protease 2 (TMPRSS2) for the spike (S) protein priming, which also leads to downregulation of ACE2 [8]. Down-regulation of ACE2 caused by Coronavirus may have a potential role in the pathogenesis of COVID-19 infection. Accordingly, people with a higher ACE/ACE2 ratio may be more at increased risk of worse Covid-19 consequences [9].

On the other hand, omega-3 fatty acids could decrease CVD risk by their anti-inflammatory anti-thrombotic function [10]. A meta-analysis comprising 15,806 patients, showed that omega-3 fatty acids associated with a 30% reduction in fatal myocardial infarction and sudden death, in addition to a 20% reduction in overall mortality [11]. To the best of our knowledge, no clinical trials have evaluated the effect of omega-3 supplementation on serum ACE/ACE2 ratio which is recently ascribed as a potential key in 2019 Covid-19 as well as CVD [5,9].

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria included males and females in the age range of 35-65 years without a medical diagnosis of COVID-19 infection.

Exclusion Criteria:

* Any subject with any chronic disease such as CVD, diabetes, or immune problems, including autoimmune diseases, chronic or severe infections was excluded.
* Pregnant, breastfeeding, and females using hormonal contraceptives were excluded.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
serum ACE levels | 10 weeks
  Angiotensin converting enzyme levels pg/mL
serum ACE2 levels | 10 weeks
  Angiotensin converting enzyme-2 levels

SECONDARY OUTCOMES:
Lipid profile mg/dL | 10 weeks
  TC,LDL,HDL,TG

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S Abu-Samak, PhD, Study Chair — Department of Clinical Pharmacy and Therapeutics , Applied Science Private University, Amman -Jordan; Sara M Daboul, MSC, Principal Investigator — Department of Clinical Pharmacy and Therapeutics , Applied Science Private University, Amman -Jordan
Locations (1):
- Mahmoud S Abu-Samak, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided